CLINICAL TRIAL: NCT03991143
Title: A Phase IIa, Placebo-controlled, Double Blind, Randomised Multicentre Pilot Study to Investigate the Efficacy, Safety and Tolerability of the Monoclonal Antibody ATH3G10 in Patients With ST-elevation Myocardial Infarction
Brief Title: Efficacy, Safety and Tolerability of ATH3G10 in Patients With ST-elevation Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Athera Biotechnologies AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATH3G10-006; 2018-003676-12 (EudraCT Number)
Record Dates: First submitted 2019-06-14; First posted 2019-06-19 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATH3G10 (Experimental): Phosphorylcholine human monoclonal antibody (ATH3G10)
  Interventions: Drug: ATH3G10
- Placebo (Placebo Comparator): Placebo to ATH3G10, 0.9% sodium chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH3G10 — intravenous
  Other Names: PC-mAB
  Arms: ATH3G10
Drug: Placebo — intravenous
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
Patients with ST-segment elevation myocardial infarction (STEMI) that have suffered a major anterior wall infarction or where coronary blood flow is less than normal in spite of successful percutaneous coronary intervention (PCI) have a poor prognosis. There are today no medical treatments that specifically reduce risk in these patients. The acute inflammatory reaction in conjunction with a STEMI and reperfusion by PCI determines the final size of the infarction and the signals leading to left ventricular remodelling.

This study is designed to assess the efficacy and safety of single intravenous injection with ATH3G10, a fully human IgG1 antibody against phosphorylcholine, in high-risk subjects with STEMI. ATH3G10 aims to reduce inflammation and thereby infarction size and remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction with ST elevation at the J-point in two contiguous leads
* Start of PCI less than 4 hours after symptom onset.

Exclusion Criteria:

* Cardiogenic chock, non-compensated acute heart failure and/or pulmonary edema.
* Previous major vascular intervention within the last 4 weeks.
* History of an infarct in the same artery that is currently affected.
* Conditions contraindicating MRI

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Left ventricular remodelling | From Visit2 (day 3) to visit 3 (day 90)
  Change in Left Ventricular End-Diastolic Volume index (LV EDVi)

SECONDARY OUTCOMES:
Myocardial Salvage index (MSi) | Visit 2 (day 3)
  Effects on myocardial salvage index (MSi) measured by MRI

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and tolerability] | From baseline (Visit 1, day 1) to visit 3 (day 90)
  Assessment of Safety and Tolerability based on incidence of AEs/SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No